CLINICAL TRIAL: NCT00228657
Title: The Formation and Severity of Pressure Ulcers Associated With 4% Albumin vs. 0.9% Sodium Chloride Administration (Substudy of SAFE Protocol 153711)
Brief Title: Formation and Severity of Pressure Ulcers Associated With 4% Albumin vs. 0.9% Sodium Chloride
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 137/99
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2005-09

CONDITIONS: Pressure Ulcer, Area; Pressure Ulcer, Grade; Albumin Level; Risk Score; Length of ICU Stay
MeSH Terms: conditions — Pressure Ulcer | interventions — Albumins; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 4% Albumin / 0.9% Sodium Chloride

SUMMARY:
Patients resuscitated with 4% Albumin will have less incidence and reduced severity of pressure injuries than patients resuscitated with 0.9% Sodium Chloride due to the improved intravascular oncotic pressure effected from higher albumin levels.

DETAILED DESCRIPTION:
Pressure ulcers incur multiple risks to the patient. The disruption of the skin is a portal of entry for infection , which may remain localised to the site or become blood borne. A pressure ulcer can lead to protein and fluid losses from the wound exudate. Many authors have theorised the existence of a relationship between the development of pressure ulcers and low serum albumin levels however, there is no strong evidence to prove this correlation. The literature does demonstrate a clear relationship between people with existing pressure ulcers and the presence of low serum albumins. Specifically serum albumin levels <30mg/dl have been associated with the incidence of pressure ulcer development.

ELIGIBILITY:
Inclusion Criteria:

Randomisation to the SAFE study -

Exclusion Criteria:

In addition to the SAFE exclusion criteria, pre-existing pressure ulcers (developed prior to ICU admission) will also be excluded-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2002-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Patients receiving 4% Albumin will have less incidence and reduced severity of pressure injuries.

SECONDARY OUTCOMES:
Is there a difference in the incidence of pressure injuries between those patients resuscitated with 4% Albumin and patients resuscitated with 0.9% Sodium Chloride
Is there a difference in the severity of pressure injuries between those patients resuscitated with 4% Albumin and patients resuscitated with 0.9% Sodium Chloride.

CONTACTS AND LOCATIONS:
Overall Officials: Shena M Graham, BN, Principal Investigator — The Alfred Hospital, Prahran, Melbourne, Australia
Locations (1):
- The Alfred Hospital, Prahran,, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Anthony D, Reynolds T, Russell L. An investigation into the use of serum albumin in pressure sore prediction. J Adv Nurs. 2000 Aug;32(2):359-65. doi: 10.1046/j.1365-2648.2000.01484.x. PMID 10964183
- [Background] Hanan K, Scheele L. Albumin vs. weight as a predictor of nutritional status and pressure ulcer development. Ostomy Wound Manage. 1991 Mar-Apr;33:22-7. No abstract available. PMID 2018614
- [Background] Cullum N, Clark M. Intrinsic factors associated with pressure sores in elderly people. J Adv Nurs. 1992 Apr;17(4):427-31. doi: 10.1111/j.1365-2648.1992.tb01926.x. PMID 1578064
- [Background] Goodrich C, March K. From ED to ICU: a focus on prevention of skin breakdown. Crit Care Nurs Q. 1992 May;15(1):1-13. doi: 10.1097/00002727-199205000-00002. No abstract available. PMID 1568151
- [Background] Peerless JR, Davies A, Klein D, Yu D. Skin complications in the intensive care unit. Clin Chest Med. 1999 Jun;20(2):453-67, x. doi: 10.1016/s0272-5231(05)70152-0. PMID 10386267
- [Background] Kuhn MM. Colloids vs crystalloids. Crit Care Nurse. 1991 May;11(5):37-44, 46-51. PMID 2026044